CLINICAL TRIAL: NCT06178536
Title: Clinical and Radiographic Assessment of a Novel Wedge Shape Implant Placed in Edentulous Narrow Ridges: Comparison of Bone Consuming and Bone Expanding Techniques for Implants Presenting Either Machined or Roughened Transcortical Portion
Brief Title: Clinical and Radiographic Assessment of a Novel Wedge Shape Implant Placed in Edentulous Narrow Ridges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Makary (Other)
Responsible Party: Sponsor-Investigator, Christian Makary, Professor, Saint-Joseph University
Organization: Saint-Joseph University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XFMD128
Record Dates: First submitted 2023-12-06; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Surgical Technique; Implant Surface

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rex implant machined transcortical portion (Experimental): Implants in these group will have a machined portion at the neck of the implant
  Interventions: Procedure: Bone Consumption; Procedure: Bone expansion
- Rex implant roughened transcortical portion (Active Comparator): Rex implants with a rough surface until the neck of the implant
  Interventions: Procedure: Bone Consumption; Procedure: Bone expansion

INTERVENTIONS:
Procedure: Bone Consumption — The surgery will be done using a bone consumption protocol
Procedure: Bone expansion — implants will be placed after a bone expansion protocol

SUMMARY:
The aim is to clinically and radiographically assess a novel wedge implant placed in narrow ridges.

* 60 wedge implants (Rex Implants, Columbus, OH, USA) will be placed using Piezosurgery® following either a bone consumption (n=30) or bone expansion technique (n=30). Each group (bone consumption and bone expansion) will be divided into 2 surface treatments: machined transcortical portion (n=15) and roughened transcortical portion (n=15).
* Record the time needed to place each implant.
* ISQ will be evaluated at Day 0, 3 weeks, 6 weeks, 3 months, 4 months, and 6 months after implant placement.
* Periapical radiographs will be performed at implant placement, loading. and 1, 3, and 5 years after loading to assess marginal bone stability.
* Buccal bone height and lingual and buccal bone thickness will be recorded post-intervention, at the time of functional loading, and at 12, 36, and 60 months after loading with CBCT.
* Digital impressions will be taken post-operatively, at loading and at 12 months after loading to monitor gingival profile.

ELIGIBILITY:
Inclusion Criteria:

1. Partially or totally edentulous patients presenting indications for a prosthetic rehabilitation supported by the upper or lower jaw implants on the basis of an accurate diagnosis and treatment planning;
2. the bone crest must be completely healed (at least six months after the loss of teeth);
3. the residual bone crest must have a width between 3 and 5 mm;
4. presence of at least 10 mm of bone height available for implant placement; 5) patient age > 18 years;

6) the patient must not wear any type of removable dentures on the treated area; 7) the patient must be capable of following the study protocol; and 8) written informed consent must be provided

Exclusion Criteria:

1. acute myocardial infarction within the last two months;
2. Uncontrolled coagulation disorders;
3. uncontrolled diabetes (HBA1c> 7.5);
4. radiation therapy to the head \ neck region in the last 24 months;
5. immunocompromised patients, HIV positive or receiving chemotherapy in the last five years;
6. past or present treatment with intravenous bisphosphonates;
7. psychological or psychiatric problems;
8. abuse of alcohol or drugs;

Ages: 35 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Implant stability | 0, 3 weeks, 6 weeks, 3 months, 4 months, and 6 months after implant placement.
  Implant stability quotient evaluation
Bone stability | At 6 months, and at 12, 36, and 60 months after loading
  Periapical radiograph and CBCT
Gingival profile monitoring | Day 0 of surgery, at 6 months and at 12 months.
  Digital impression superimposition

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No